CLINICAL TRIAL: NCT00982787
Title: A Phase II Randomized, Placebo Controlled, Double-blind, Cross-over Clinical Trial to Test the Safety and Potential Anticonvulsant Efficacy of a Botanical Extract From Passiflora Incarnata, in Patients With Partial Onset Epilepsy.
Brief Title: Safety and Anticonvulsant Efficacy of Passiflora Incarnata Extract in Patients With Partial Epilepsy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Oregon Clinical and Translational Research Institute (Other); Oregon's Wild Harvest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 3107; 5K23AT001933-03 (NIH)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Partial Epilepsy
Keywords: Epilepsy; Seizures; Passiflora
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Botanical extract from Passiflora incarnata
- 2 (Placebo Comparator)
  Interventions: Drug: Botanical extract from Passiflora incarnata

INTERVENTIONS:
Drug: Botanical extract from Passiflora incarnata — Dosage form: Liquid Passiflora extract
  Dosage: 10ml (equivalent of 2.2 g of dried Passiflora)
  Frequency: Once/Twice a day
  Duration: 11 week intervention period
  Other Names: Whole ethanolic extract from Passiflora Incarnata dried herb

SUMMARY:
The purpose of the Phase II clinical trial will be to see if a botanical extract from the plant Passiflora incarnata can improve seizure control and reduce anxiety in patients diagnosed with partial epilepsy.

The investigators will randomize approximately 25 participants with partial epilepsy for this placebo controlled, double blind, and crossover study. All patients will be scheduled for 10 clinic visits and four telephone visits during the 32-week period of the trial. After enrollment into the study, all participants will begin a 9-week observation phase, which serves as an individual baseline control. After 9 weeks participants will be randomized to receive either study drug or placebo for an 11 week study period. After completion of the 11 week study period, patients will crossover to the other study drug/placebo arm for another 11 weeks. Epilepsy participants will continue taking their anti-epileptic medication as currently prescribed. The investigators will find participants through the OHSU clinics, by notifying local neurologists, anthroposophical and naturopathic practices, and by advertising the study via the local chapter of the American Epilepsy Society.

Routine blood tests, physical examinations and tests to monitor heart, brain and muscle activities will screen for any adverse effects. The primary outcome measure will be seizure frequency through seizure diaries. Attention and performance tests, neurological and quality of life questionnaires will be completed to assess the secondary outcome measures of anxiety, cognitive function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old.
* Reliable history of seizure semiology, EEG or EEG video telemetry confirming the diagnosis of partial epilepsy.
* Seizure frequency of at least 6 complex partial seizures over the 9 weeks prior to enrollment, with no 3 week period with less than one seizure, in spite of adequate treatment with a stable anticonvulsant dosage with one or two anticonvulsants for at least one month. Every seizure in a cluster will count as a separate seizure.
* Willing to maintain current anticonvulsant dosage for 32 weeks. Tapering off a third anticonvulsant up to one month prior to enrollment to allow study participation is permitted. Consent will be obtained prior to tapering of a third anticonvulsant. Habitual use of an additional rescue medication such as lorazepam for excess seizure activity is permitted but not more frequently than once every three weeks.
* Women of childbearing potential need to have a negative urine pregnancy test and practice two simultaneous methods of birth control, which may not include oral contraceptives. Due to drug interactions, oral contraceptives are not considered a safe method of birth control in patients using anticonvulsant medications. Women who are at least two years post-menopausal will be exempt from the pregnancy test or birth control requirements.

Exclusion criteria:

* Unreliable history of seizure semiology.
* Seizure frequency less than six complex partial seizures over 9 weeks or no seizure in any 3-week period in the 9 weeks prior to enrollment.
* Patients in whom it is anticipated that current standard of care would mandate a change in their conventional epilepsy treatment during the time period of the study will be excluded.
* Patients with a widely fluctuating seizure frequency (good months and bad months) or a history of status epilepsy will be excluded.
* Women who are currently pregnant or lactating
* Patients with other serious medical problems, such as brain tumors, cancer, stroke, significant heart disease or psychiatric disorders such as schizophrenia or major depression will be excluded.
* Patients with progressive epilepsy syndromes, neurodegenerative disorders or dementia will be excluded.
* Patients with impaired renal or hepatic function as detected by abnormal BUN or AST/ALT/alk phos on initial screening will be excluded.
* Patients at increased risk for ventricular arrhythmias (history of heart failure, prolonged QTc > 450 ms, family history of prolonged QT syndrome, hypokalemia, or those using any diuretics or drugs which prolong the QT, see http://www.azcert.org) will be excluded.
* Patients with a high likelihood of psychogenic or non-epileptic seizures will be excluded by the following method previously developed at the Oregon Health and Science University (OHSU) epilepsy program.
* Patients who use alcohol, drugs or have participated in another clinical trial in the past 6 months, and patients who are found to be less than 80% compliant with their documentation of seizure and medication diary will be excluded as will patients unwilling to stop using oral contraceptives at the time of study enrollment. Patients who agree to participate and are currently taking botanicals will be asked to discontinue them at enrollment, as these may confound study results or cause safety issues.
* Patients who are found to have generalized spike and wave discharges, diagnostic of primary generalized epilepsy, on their EEG will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency | 32 weeks

SECONDARY OUTCOMES:
Anxiety, sedation, quality of life | 32 weeks
Cognitive testing | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Siegward M Elsas, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science Universtiy, Portland, Oregon, United States